CLINICAL TRIAL: NCT02020005
Title: Evaluation of Cessation Preferences of Menthol Smokers
Brief Title: Evaluation of Cessation Preferences of Menthol Smoker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2013NTLS014; NCT01978197 (obsolete NCT alias)
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Smoking Cessation
Keywords: menthol cigarettes; smoking cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Chewing Gum

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- non-flavored 2mg nicotine gum (Experimental): All subjects will test six different nicotine replacement products over the course of the 2-week product sampling phase. The six nicotine replacement products being tested are non-flavored 2mg nicotine gum, non-flavored 4mg nicotine gum, mint-flavored 2mg nicotine gum, mint-flavored 4mg nicotine gum, non-flavored nicotine inhaler and mint-flavored inhaler. The order in which the subjects test these products will be randomized and subjects will be blinded to the nicotine content of the product but will be instructed about the flavor of the product.
  Interventions: Other: Non-flavored 2mg nicotine gum
- non-flavored 4mg nicotine gum (Experimental): All subjects will test six different nicotine replacement products over the course of the 2-week product sampling phase. The six nicotine replacement products being tested are non-flavored 2mg nicotine gum, non-flavored 4mg nicotine gum, mint-flavored 2mg nicotine gum, mint-flavored 4mg nicotine gum, non-flavored nicotine inhaler and mint-flavored inhaler. The order in which the subjects test these products will be randomized and subjects will be blinded to the nicotine content of the product but will be instructed about the flavor of the product.
  Interventions: Other: Non-flavored 4mg nicotine gum
- mint-flavored 2mg nicotine gum (Experimental): All subjects will test six different nicotine replacement products over the course of the 2-week product sampling phase. The six nicotine replacement products being tested are non-flavored 2mg nicotine gum, non-flavored 4mg nicotine gum, mint-flavored 2mg nicotine gum, mint-flavored 4mg nicotine gum, non-flavored nicotine inhaler and mint-flavored inhaler. The order in which the subjects test these products will be randomized and subjects will be blinded to the nicotine content of the product but will be instructed about the flavor of the product.
  Interventions: Other: Mint-flavored 2mg nicotine gum
- mint-flavored 4mg nicotine gum (Experimental): All subjects will test six different nicotine replacement products over the course of the 2-week product sampling phase. The six nicotine replacement products being tested are non-flavored 2mg nicotine gum, non-flavored 4mg nicotine gum, mint-flavored 2mg nicotine gum, mint-flavored 4mg nicotine gum, non-flavored nicotine inhaler and mint-flavored inhaler. The order in which the subjects test these products will be randomized and subjects will be blinded to the nicotine content of the product but will be instructed about the flavor of the product.
  Interventions: Other: Mint-flavored 4mg nicotine gum
- non-flavored nicotine inhaler (Experimental): All subjects will test six different nicotine replacement products over the course of the 2-week product sampling phase. The six nicotine replacement products being tested are non-flavored 2mg nicotine gum, non-flavored 4mg nicotine gum, mint-flavored 2mg nicotine gum, mint-flavored 4mg nicotine gum, non-flavored nicotine inhaler and mint-flavored inhaler. The order in which the subjects test these products will be randomized and subjects will be blinded to the nicotine content of the product but will be instructed about the flavor of the product.
  Interventions: Other: Non-flavored nicotine inhaler
- mint-flavored inhaler (Experimental): All subjects will test six different nicotine replacement products over the course of the 2-week product sampling phase. The six nicotine replacement products being tested are non-flavored 2mg nicotine gum, non-flavored 4mg nicotine gum, mint-flavored 2mg nicotine gum, mint-flavored 4mg nicotine gum, non-flavored nicotine inhaler and mint-flavored inhaler. The order in which the subjects test these products will be randomized and subjects will be blinded to the nicotine content of the product but will be instructed about the flavor of the product.
  Interventions: Other: Mint-flavored nicotine ihaler

INTERVENTIONS:
Other: Non-flavored 2mg nicotine gum
  Arms: non-flavored 2mg nicotine gum
Other: Non-flavored 4mg nicotine gum
  Arms: non-flavored 4mg nicotine gum
Other: Mint-flavored 2mg nicotine gum
  Arms: mint-flavored 2mg nicotine gum
Other: Mint-flavored 4mg nicotine gum
  Arms: mint-flavored 4mg nicotine gum
Other: Non-flavored nicotine inhaler
  Arms: non-flavored nicotine inhaler
Other: Mint-flavored nicotine ihaler
  Arms: mint-flavored inhaler

SUMMARY:
The primary aim of this study is to determine menthol smokers' perception, product preference, and pattern of use across six products including, mint-flavored nicotine gum; non-flavored nicotine gum; mentholated nicotine inhaler; and non-menthol nicotine inhaler. Participants will undergo an orientation and baseline assessment followed by a 2-week product sampling phase. At the end of the 2 weeks of sampling, subjects will select a product to use during the following 2-week smoking cessation phase. This 2-week abstinence phase is followed by one week of abrupt withdrawal of the product. This study design was successfully used in a study we conducted that examined the smokers' preference for a variety or oral tobacco products.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as African American or Black;
* Aged 18 years or older;
* High school graduate or GED;
* Smoking at least 10 cigarettes daily for the past year;
* Usually smoked mentholated cigarette brand (greater than 80% of the time) in the past two years;
* Good physical health (no unstable medical condition);
* No contraindications for nicotine inhaler or gum use, such as mouth sores or significant dental or jaw problems;
* Stable, good health.

Exclusion Criteria:

* Recent unstable or untreated psychiatric diagnosis including substance abuse, as determined by the DSM-IV criteria;
* Currently using other tobacco or nicotine products other than cigarettes;
* Pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Product preference for nicotine replacement | 6 weeks
  To determine menthol smokers' product perception and preference across 6 different types of products with varying mint content.

SECONDARY OUTCOMES:
Nicotine content preference | 6 weeks
  To determine menthol smokers' product perception and preference across 6 different types of products with varying nicotine content.

CONTACTS AND LOCATIONS:
Overall Officials: Kola Okuyemi, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota, United States